CLINICAL TRIAL: NCT01948609
Title: Prospective Research of Outcomes After Salpingo-oophorectomy
Acronym: PROSper
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 13-11221
Record Dates: First submitted 2013-09-12; First posted 2013-09-23 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: BRCA1 Gene Mutation; BRCA2 Gene Mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood; serum; EDTA Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated with RRSO: Women with the BRCA gene 1/2 mutation who choose to undergo risk reducing salpingo-oophorectomy (RRSO) treatment.
- No RRSO treatment: Women with the BRCA gene 1/2 mutation who choose non-surgical treatment.

SUMMARY:
PROSper is a prospective cohort study of 100 women 35-50 years of age with BRCA 1/2 mutations who have elected to either undergo risk reducing salpingo-oophorectomy (RRSO) or nonsurgical management. The investigators will compare the change in cardiovascular health, bone health, sexual function, quality of life, and menopausal symptoms over 3 years of follow-up between women who undergo RRSO (baseline just prior to surgery) and age-matched controls that do not undergo RRSO.

The investigators hypothesis is that women who undergo a premature surgical menopause induced by RRSO have worse cardiovascular health and bone health compared with women who do not undergo RRSO.

ELIGIBILITY:
Inclusion Criteria:

* BRCA mutation 1/2 or "Variant suspected deleterious" mutation.
* Female
* Age 35-50 years
* Able to undergo RRSO
* Speaks English
* Able to give informed consent

Exclusion Criteria:

* Prior history of bilateral oophorectomy
* BRCA 1/2 deleterious mutation
* Plans to move out of geographic region in next 3 years
* Unable to travel to study visits

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study participants will be women 35-50 years old with a confirmed diagnosis of a deleterious BRCA 1/2 mutation recruited through UCSF.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in risk of cardiovascular disease and osteoporosis at 36 months. | Baseline to 36 Months
  We will use dual-energy x-ray absorptiometry (DEXA) scan results and Intima-media thickness of the carotid artery (IMT) testing to assess changes in bone mineral density and carotid artery intima media thickness, respectively.
Change in baseline sexual functioning and quality of life at 36 months. | Baseline to 36 Months
  We will use standard questionnaires to assess changes in overall quality of life and sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jacoby, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan LN, Chen LM, Goldman M, Mak JS, Bauer DC, Boscardin J, Schembri M, Bae-Jump V, Friedman S, Jacoby VL. Changes in Bone Density in Carriers of BRCA1 and BRCA2 Pathogenic Variants After Salpingo-Oophorectomy. Obstet Gynecol. 2023 Jul 1;142(1):160-169. doi: 10.1097/AOG.0000000000005236. Epub 2023 Jun 7. PMID 37290104
- See also: BRCA 1 Studies at UCSF — https://clinicaltrials.ucsf.edu/brca-1-gene-mutation
- See also: BRCA 2 Studies at UCSF — https://clinicaltrials.ucsf.edu/brca-2-gene-mutation